CLINICAL TRIAL: NCT04924101
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Pembrolizumab Plus Investigational Agents in Combination With Etoposide and Cisplatin or Carboplatin for the First-Line Treatment of Participants With Extensive-Stage Small Cell Lung Cancer (KEYNOTE-B99)
Brief Title: Efficacy and Safety of Pembrolizumab Plus Investigational Agents in Combination With Chemotherapy as First-Line Treatment in Extensive-Stage Small Cell Lung Cancer (ES-SCLC) (MK-3475-B99/ KEYNOTE-B99)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B99; MK-3475-B99 (Other: MSD); KEYNOTE-B99 (Other: MSD); 2023-506538-56-00 (Registry Identifier: EU CT); U1111-1293-9965 (Registry Identifier: UTN)
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Death-Ligand 2 (PDL2, PD-L2); Pembrolizumab (MK-3475)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Etoposide; etoposide phosphate; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + MK-4830 + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg IV infusion on Day 1 of each cycle (cycle length = 3 weeks) every 3 weeks (Q3W) up to 35 administrations (up to approximately 2 years) or until disease progression (PD) or discontinuation, MK-4830 800 mg IV infusion on Day 1 of each cycle Q3W, up to 35 administrations (up to approximately 2 years) or until PD or discontinuation; etoposide 100 mg/m^2 on Days 1, 2, 3 of each cycle for up to 4 cycles (up to approximately 12 weeks) and cisplatin 75 mg/m^2 or carboplatin AUC 5 mg/ml/min IV, Day 1 of each cycle Q3W up to 4 cycles (up to approximately 12 weeks) or until PD or discontinuation.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin
- Pembrolizumab + Boserolimab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg IV infusion on Day 1 of each cycle Q3W up to 35 administrations (up to approximately 2 years) or until PD or discontinuation, boserolimab 30 mg IV infusion on Day 1 of each cycle (cycle length = 6 weeks) every 6 weeks (Q6W), up to 18 administrations (up to approximately 2 years) or until PD or discontinuation; etoposide 100 mg/m^2 on Days 1, 2, 3 of each cycle for up to 4 cycles (up to approximately 12 weeks) and cisplatin 75 mg/m^2 or carboplatin AUC 5 mg/ml/min IV, Day 1 of each cycle Q3W up to 4 cycles (up to approximately 12 weeks) or until PD or discontinuation.
  Interventions: Biological: Pembrolizumab; Biological: Boserolimab; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin
- Pembrolizumab + Lenvatinib + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg IV infusion on Day 1 of each 3 week cycle (Q3W) up to 35 administrations (up to approximately 2 years) or until PD or discontinuation, lenvatinib 8 mg once daily (QD) orally up to Cycles 1-4 cycles and up to 20 mg QD orally for Cycles 5-31 or until PD or discontinuation; etoposide 100 mg/m^2 on Days 1, 2, 3 of each cycle for up to 4 cycles (up to approximately 12 weeks) and cisplatin 75 mg/m^2 or carboplatin AUC 5 mg/ml/min IV, Day 1 of each cycle Q3W up to 4 cycles (up to approximately 12 weeks) or until PD or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
Biological: MK-4830 — IV infusion
  Arms: Pembrolizumab + MK-4830 + Chemotherapy
Biological: Boserolimab — IV infusion
  Other Names: MK-5890
  Arms: Pembrolizumab + Boserolimab + Chemotherapy
Drug: Lenvatinib — Oral capsule
  Other Names: LENVIMA®; KISPLYX®; MK-7902; E7080
  Arms: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: Etoposide — IV infusion
  Other Names: Etopophos®; Vepesid®; Toposar®; VP-16; Etoposide phosphate
Drug: Cisplatin — IV infusion
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Carboplatin — IV infusion
  Other Names: Paraplatin; Paraplatin NovaPlus; Carboplatin N+ Novaplus; Carboplatin Novaplus; PremierPro Rx Carboplatin

SUMMARY:
The purpose of this study is to evaluate the use of investigational agents (MK-4830, boserolimab (MK-5890) and lenvatinib (MK-7902)) in combination with pembrolizumab (MK-3475) and etoposide/platinum chemotherapy for the first-line treatment of participants with extensive-stage small cell Lung Cancer (ES-SCLC). No formal hypothesis testing will be performed for this study.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of extensive-stage small cell lung cancer (ES-SCLC) in need of first-line therapy
* Has ES-SCLC defined as Stage IV (T any, N any, M1a/b/c) by the American Joint Committee on Cancer, Eighth Edition
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception for each study intervention is as follows: Lenvatinib (7 days); Etoposide, Cisplatin, or Carboplatin (180 days) and Pembrolizumab, MK-4830, or (no contraception measures); refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent or must agree to use contraception per protocol unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman/women of childbearing potential (WOCBP) or is a WOCBP and uses a contraceptive method that is highly effective with low user dependency or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention and agrees not to donate eggs to others or freeze/store for her own use for the purpose of reproduction during this period. The length of time required to continue contraception for each study intervention is as follows: Lenvatinib (30 days), Etoposide, Cisplatin, or Carboplatin (180 days), and Pembrolizumab, MK-4830, or Boserolimab (120 days)
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours (urine test) or 72 hours (serum test) before the first dose of study intervention
* Abstains from breastfeeding during the study intervention period and for at least 120 days after study intervention
* Has measurable disease per RECIST 1.1 as assessed by local site investigator/radiology and verified by blinded independent central review (BICR)
* Submits an archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated where such sample exist
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days before randomization
* Has adequate organ function within 10 days before the first dose of study intervention
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg with no changes in antihypertensive medications within 1 week before randomization

Exclusion Criteria:

* Has had major surgery within 3 weeks before first dose of study interventions
* Has a preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
* Has urine protein ≥1 g/24 hours
* Has a left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multiple gated acquisition (MUGA) or echocardiogram (ECHO)
* Prolongation of QT interval with Fridericia's correction (QTcF) interval to >480 ms
* Has clinically significant cardiovascular disease or major arterial thromboembolic event within 12 months before first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has active hemoptysis within 3 weeks before the first dose of study intervention
* Has gastrointestinal malabsorption or any other condition that might affect oral study intervention absorption
* Has serious nonhealing wound, ulcer, or bone fracture within 28 days before first dose of study intervention
* Has any major hemorrhage or venous thromboembolic events within 3 months before the first dose of study intervention. Participants with venous thrombosis diagnosed more than 3 months before the first dose of study intervention must be on stable doses of anticoagulants
* Has a history of inflammatory bowel disease
* Has a history of a gastrointestinal perforation within 6 months before the first dose of study intervention
* Is considered a poor medical risk due to a serious, uncontrolled medical disorder or nonmalignant systemic disease
* Has received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received prior treatment (chemotherapy, radiotherapy, or surgical resection) including investigational agents for SCLC
* Is expected to require any other form of antineoplastic therapy for SCLC, including radiation therapy, while on study
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation. A participant that meets this exclusion criterion but is otherwise deemed eligible for the study may be randomized across the specific intervention groups.
* Has symptomatic ascites, pleural effusion, or pericardial effusion. A participant who is clinically stable following treatment for these conditions is eligible
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with brain metastases may participate only if they satisfy all of the following: a) Completed treatment at least 14 days before the first dose of study intervention b) Have no evidence of new or enlarging brain metastases confirmed by posttreatment repeat brain imaging performed at least 4 weeks after pretreatment brain imaging, and c) Are neurologically stable without the need for steroids for at least 7 days before the first dose of study intervention as per local site assessment. Participants with untreated brain metastases will be allowed if they are asymptomatic, the investigator determines there is no immediate CNS-specific treatment required, there is no significant surrounding edema, and the brain metastases are of 5 mm or less in size and 3 or fewer in number
* Has a history of severe hypersensitivity reaction to any study intervention and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a known history of, or active, neurologic paraneoplastic syndrome
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection and/or Hepatitis B virus infection or an active Hepatitis C infection
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 5 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Six-Month Progression-Free Survival (PFS) as Assessed by BICR per RECIST 1.1 | Up to approximately 6 months
  Six-month PFS is defined as the survival without documented disease progression (PD) per RECIST 1.1 by BICR or death due to any cause, whichever occurs first at 6 months after randomization. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) as Assessed by BICR per RECIST 1.1 | Up to approximately 5 years
  DOR is defined as the time from first documented evidence of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) until first documented PD per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) as Assessed by BICR per RECIST 1.1 | Up to approximately 5 years
  PFS is defined as the time from randomization to the first documented PD per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Percent Change From Baseline in Tumor Size as Assessed by BICR | Baseline, 5 years
  Tumor size change is defined as the percent change from baseline in the sum of the diameters of the target lesions as assessed by BICR. Percent change from baseline in tumor size as assessed by BICR will be presented.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be presented.
Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) Global Health Status/Quality of Life Scale (Items 29 and 30) at Week 19 | Baseline, Week 19
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The mean change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (49):
- United States (14):
  - Banner MD Anderson Cancer Center ( Site 0102), Gilbert, Arizona
  - University of Colorado Anschutz Medical Campus ( Site 0104), Aurora, Colorado
  - Georgia Cancer Specialists ( Site 0106), Atlanta, Georgia
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0130), Fort Wayne, Indiana
  - Baptist Health Lexington-Research ( Site 0108), Lexington, Kentucky
  - MFSMC-HJWCI-Oncology Research ( Site 0128), Baltimore, Maryland
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0122), Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0129), Omaha, Nebraska
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0114), Mineola, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0115), New York, New York
  - Cleveland Clinic-Taussig Cancer Center ( Site 0116), Cleveland, Ohio
  - UPMC Hillman Cancer Center ( Site 0127), Pittsburgh, Pennsylvania
  - St Francis Cancer Center-Research Office ( Site 0117), Greenville, South Carolina
  - Virginia Cancer Institute ( Site 0119), Richmond, Virginia
- Austria (2):
  - Klinik Penzing-2. Lungenabteilung ( Site 2101), Vienna, Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 2100), Vienna
- Canada (3):
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 2003), Hamilton, Ontario
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 2005), Kingston, Ontario
  - St. Marys Hospital Center ( Site 2000), Montreal, Quebec
- Hungary (5):
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 2800), Szolnok, Jász-Nagykun-Szolnok
  - Országos Korányi Pulmonológiai Intézet-XIV. Tüdöbelgyógyászat ( Site 2806), Budapest, Pest County
  - Torokbalint Tudogyogyintezet-Onkopulmonologiai Jarobeteg Centrum ( Site 2801), Törökbálint, Pest County
  - Zala Megyei Szent Rafael Kórház-Pulmonológia ( Site 2805), Zalaegerszeg, Zala County
  - Semmelweis University-Pulmonológiai Klinika ( Site 2802), Budapest
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 2600), Haifa
  - Shaare Zedek Medical Center ( Site 2602), Jerusalem
  - Meir Medical Center ( Site 2601), Kfar Saba
  - Rabin Medical Center-Oncology ( Site 2604), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 2603), Ramat Gan
- Italy (3):
  - Ospedale San Raffaele-Oncologia Medica ( Site 2303), Milan, Lombardy
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica ( Site 2300), Siena, Tuscany
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Toracica ( Site 2304), Milan
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Zespó Grulicy i Chorób Puc w Olsztynie-Oddzial Onkologii z Pododdzialem Chemi, Olsztyn, Warmian-Masurian Voivodeship
- Russia (4):
  - Krasnoyarsk Regional Oncology Dispensary, Named after Krizhanovsky ( Site 2708), Krasnoyarsk, Krasnoyarsk Krai
  - GBUZ "SPb CRPCstmc(o)" ( Site 2705), Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology-Department of Chemotherapy and Innovative Technologies ( S, Saint Petersburg, Sankt-Peterburg
  - Scientific research institution of oncology named after N.N. Petrov-Thoracic oncology ( Site 2704), Saint Petersburg
- South Korea (7):
  - Seoul National University Bundang Hospital ( Site 1104), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital ( Site 1106), Suwon, Kyonggi-do
  - Chungbuk National University Hospital ( Site 1107), Cheongju-si, North Chungcheong
  - Seoul National University Hospital ( Site 1101), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1105), Seoul
  - Asan Medical Center-Department of Oncology ( Site 1103), Seoul
  - Samsung Medical Center ( Site 1100), Seoul
- Spain (3):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals ( Site 2403), L'Hospitalet de Llobregat, Catalonia
  - Hospital Insular de Gran Canaria ( Site 2402), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 2401), Barcelona
- Cantonal Hospital St.Gallen-Oncology & Hematology ( Site 2502), Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26259&tenant=MT_MSD_9011